CLINICAL TRIAL: NCT00924755
Title: Early Outcome of Inguinal Hernia Repair With Biomerix Surgical Mesh Using the Lichtenstein Technique
Brief Title: Study of Surgical Mesh for Inguinal Hernia Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biomerix (Industry)
Responsible Party: Christina Kichula, Biomerix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMX-2008-03
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Hernia, Inguinal
Keywords: Surgical mesh
MeSH Terms: conditions — Hernia, Inguinal | interventions — Surgical Mesh

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Biomerix Revive™ (surgical mesh for inguinal hernia repair) — Inguinal hernia repair using a tension-free onlay patch, Lichtenstein-style.
  Other Names: Revive

SUMMARY:
The purpose of this study is to assess the early outcomes when using the Biomerix Revive™ as a tension-free onlay patch, Lichtenstein-style, in patients who are candidates for primary, unilateral, open inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* male ≥19 years old
* symptomatic and palpable inguinal hernia
* candidate for unilateral, primary, open inguinal hernia repair using the Lichtenstein technique
* will comply with required follow-up study visits
* willing and able to provide written informed consent

Exclusion Criteria:

* BMI ≥35
* life expectancy of <3 years
* strangulated hernia
* urologic disorder and/or previous urologic surgery in the testicular area (with the exception of prostate surgery)
* active abdominal surgical condition such as bowel obstruction or perforation
* local or systemic infection or peritonitis
* known disease that impairs wound healing
* anti-platelet therapy (other than aspirin) for >7 days preceding the surgical procedure
* previous ipsilateral groin incision
* receiving immunosuppressive therapy and/or has undergone radiation therapy to the affected groin area
* uncontrolled insulin-dependent diabetic with Hgb1Ac greater than 8
* advanced cirrhosis with Child-Turcott Class of C or higher
* severe COPD requiring home oxygen
* diagnosed with chronic pain syndrome or is undergoing treatment for pain management
* candidate for another major surgical procedure with the inguinal hernia repair
* enrolled in another investigational study that may confound the results of this study
* known drug abuser
* on anti-psychotic medications
* Worker's Compensation case

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-10 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Technical success with no complications through 6 weeks. | 6 weeks

SECONDARY OUTCOMES:
Hernia recurrence | 1 year
Pain and functional status | 10 day, 6 weeks, 6 months 1 year
Incidence of complications | 10 days, 6 weeks, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Samir S Awad, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Creighton University, Omaha, Nebraska
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas